CLINICAL TRIAL: NCT07340814
Title: A Long-term Follow-up Study of Patients Who Received MB-105
Status: Not yet recruiting | Type: Observational
Sponsor: March Biosciences Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: MB-105-202
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Any Patient Treated With MB-105

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Open Observation: All patients who previously received MB-105 on another study
  Interventions: Biological: MB-105

INTERVENTIONS:
Biological: MB-105 — This is an observational study with no study product administered because it is the LTFU study for patients who received the product in another study

SUMMARY:
This study is to fulfil the regulatory requirement for 15-year follow-up for patients treated with MB-105 in any study

DETAILED DESCRIPTION:
This study is for long term follow up of efficacy and safety for any patient treated with MB-105 who has consented to joining the LTFU study. There are no exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

Received MB-105 Signed informed consent Agree to transfer of samples from previous study Able to comply with study requirements

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who previously received MB-105 and consent to participate
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-02-27 (Estimated); Primary Completion 2040-10-15 (Estimated); Study Completion 2040-10-15 (Estimated)

PRIMARY OUTCOMES:
Assess long term safety of MB-105 in patients who received MB-105 | 15 Years
  SAEs

SECONDARY OUTCOMES:
Assess long term efficacy of MB-105 in patients who received MB-105 | 15 Years
  Time to progression/relapse in those who have not yet relapsed and overall survival

IPD SHARING:
Plan to Share IPD: Undecided